CLINICAL TRIAL: NCT03692832
Title: Laparoscopic Versus Vaginal Hysterectomy for Benign Gynaecological Disease in Ain Shams University Maternity Hospital: A Randomized Clinical Trial
Brief Title: Laparoscopic vs Vaginal Hysterectomy for Benign Gynaecological Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hamdy Bakry Alqenawy, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LH-VH
Record Dates: First submitted 2018-09-10; First posted 2018-10-02 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Benign Gynecological Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Experimental): 40 patients undergoing laparoscopic hysterectomy
  Interventions: Procedure: LH
- Group V (Active Comparator): 40 patients undergoing vaginal hysterectomy
  Interventions: Procedure: VH

INTERVENTIONS:
Procedure: LH — Laparoscopic hysterectomy following AAGL class IV E, vault closed vaginally
  Arms: Group L
Procedure: VH — Vaginal hysterectomy following Heaney technique
  Arms: Group V

SUMMARY:
This study is designed to compare laparoscopic and vaginal hysterectomy in women with benign gynaecological disease in Ain Shams University Maternity Hospital.

DETAILED DESCRIPTION:
The current trial evaluates the performance and short-term postoperative outcomes of these two approaches for hysterectomy in Ain Shams University Maternity Hospital, a major tertiary hospital in Greater Cairo, and one of Egypt's leading centers in terms of provision of public medical service.

Eighty patients with benign indications, with no contraindications to neither laparoscopic nor vaginal approaches, were randomized into two equal groups, to undergo either of the two procedures: LH or VH.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing hysterectomy for benign gynaecological disease (e.g., dysfunctional uterine bleeding, adenomyosis, fibroids).

Exclusion Criteria: Women with:

* known tubo-ovarian pathology requiring primary laparotomy, e.g. large adnexal masses
* known neoplasia requiring pelvic lymphadenectomy
* pelvic organ prolapse requiring additional procedures, e.g., uterine procidentia (complete prolapse), enterocoele
* conditions interfering with laparoscopic surgery, e.g. cardio-pulmonary disease, obesity (BMI 30 kg/m2 or more)
* large uteri interfering with vaginal hysterectomy (size >16 gestational weeks)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Operative time | duration of surgical procedure
  Total operative time (minutes) for LH versus VH; from introduction of the first laparoscopy port or vaginal incision, till suturing the vaginal vault.

SECONDARY OUTCOMES:
Blood loss | intra-operative
  Blood loss (mL): by measuring suctioned blood (subtracting irrigation volumes), Weighing sponges (weight difference of soaked and dry surgical gauzes, 1 g ≃ 1 mL), or according to Gross (1983) formula (mL)
Blood transfusion | 24 hours post-operative
  Need for blood transfusion
Proportion of successful vaginal opportunistic salpingectomy | intra-operative
  Proportion of patients with successful vaginal opportunistic salpingectomy or salpingo-oophorectomy compared to laparoscopic approach, and factors for non completion
Surgical complications | intra-operative
  Surgical complications: visceral or vascular injuries, vaginal cuff haematoma or dehiscence
Post-operative pain assessed using visual analogue scale for pain intensity | first 24 hours post-operative
  Post-operative pain: assessed using visual analogue scale for pain intensity at 2, 6 and 24 hours post-operative
Febrile morbidity | first 24 hours post-operative
  Post-operative fever (temperature assessed in degrees Celsius)
Change in serum markers for inflammation | first 24 hours post-operative
  Inflammatory response serum markers compared pre- and 24-h postoperatively (e.g. C-reactive protein or interleukin-6 according to availability)
Hospital-stay | 1 week
  Post-operative hospital-stay (hours)
Healthcare costs | 1 week
  Healthcare costs (EGP), including consumables, medications, and admission fees.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Faculty of Medicine, Cairo, Egypt